CLINICAL TRIAL: NCT00033189
Title: An Open-label Pilot Study of Coenzyme Q10 in Steroid-Treated Duchenne Muscular Dystrophy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cooperative International Neuromuscular Research Group (Network)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNMC0301
Record Dates: First submitted 2002-04-08; First posted 2002-04-09 (Estimated); Last update posted 2010-11-16 (Estimated); Status verified 2010-11

CONDITIONS: Muscular Dystrophy, Duchenne
Keywords: duchenne; dystrophy; DMD; clinical trial; CINRG
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — coenzyme Q10

INTERVENTIONS:
Drug: Coenzyme Q10

SUMMARY:
This study will help to determine the safety and efficacy of the nutritional supplement Coenzyme Q10 when added to steroids as a treatment for Duchenne muscular dystrophy (DMD). Boys with DMD who are enrolled in this study will should be on a stable dose of steroids for at least six months, and will remain on their usual dose throughout the study. They will complete two screening visits within a one-week period, and if enrolled will then have their strength tested monthly for three months before beginning therapy with Coenzyme Q10. Once Coenzyme Q10 therapy is started, participants will have their strength tested monthly for six months. Following the six month treatment period, participants will be given the option to remain on Coenzyme Q10 until the study is completed.

ELIGIBILITY:
Subject Inclusion Criteria

1. Age: 5 - 11 years old
2. Ambulant
3. Diagnosis of DMD confirmed by at least one the following:

   * Positive X-linked family history for typical Duchenne muscular dystrophy in older male relatives (onset by age 5 yr., wheelchair-bound by age 12 yr.) OR
   * Dystrophin immunofluorescence and/or immunoblot showing complete dystrophin deficiency, and clinical picture consistent with typical Duchenne dystrophy OR
   * Gene deletion test positive (missing one or more exons) in the central rod domain (exons 25-60) of dystrophin, where reading frame can be predicted as 'out-of-frame', and clinical picture consistent with typical Duchenne dystrophy.
4. On Glucocorticosteroids: Children must be on a steady dose of prednisone or deflazacort, on any schedule (Daily, alternate days, 10 days on, 10 days off or twice a week), for the last 6 months before starting the clinical trial. Dose of steroid or schedule cannot be altered during the study.
5. Evidence of muscle weakness by MRC score or clinical functional evaluation
6. Ability to provide reproducible repeat QMT bicep score within 10% of first assessment score.
7. Ability to swallow tablets

Subject Exclusion Criteria

1. Failure to achieve one or more of the diagnostic inclusion criteria cited above.
2. Symptomatic DMD carrier
3. Previous (6 months or less) or current use of Coenzyme Q10 (for DMD or any other disease)
4. Use of carnitine, other amino acids, creatine, glutamine, or any herbal medicines within the last 3 months.
5. History of significant concomitant illness or significant impairment of renal or hepatic function.

Ages: 5 Years to 11 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15
Dates: Start 2001-09; Study Completion 2005-01

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Washington University-St. Louis, St Louis, Missouri